CLINICAL TRIAL: NCT03063398
Title: PAPPEI: Post Acute Pancreatitis Pancreatic Exocrine Insufficiency
Brief Title: Post Acute Pancreatitis Pancreatic Exocrine Insufficiency
Acronym: PAPPEI
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, George Papachristou, Principal Investigator, Ohio State University
Other Study IDs: STUDY19080096
Record Dates: First submitted 2017-02-02; First posted 2017-02-24 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and fecal samples will be collected for future Pancreatitis studies concerning EPI or genetics.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients after acute pancreatitis: Such patients will be followed and assessed for the development of Exocrine Pancreatic Insufficiency. 'No intervention, this is an observational study.
  Interventions: Diagnostic Test: No intervention, this is an observational study

INTERVENTIONS:
Diagnostic Test: No intervention, this is an observational study — Assessment for exocrine pancreatic insufficiency

SUMMARY:
This study is a proposed a comprehensive prospective assessment of exocrine pancreatic insufficiency (EPI), nutritional status, and quality of life (QOL) during the early re-feeding phase, at 3 months, and 12 months following an AP attack.

DETAILED DESCRIPTION:
This study is a proposed a comprehensive prospective assessment of exocrine pancreatic insufficiency (EPI), nutritional status, and quality of life (QOL) during the early re-feeding phase, at 3 months, and 12 months following an AP attack. A blood sample will be collected for measurement of nutritional markers and a fecal sample for elastase-1, and data regarding demographics, etiology, history of previous pancreatitis episodes, and their hospital course (imaging findings, interventions, length of stay, intensive care admission, and severity based on the Revised Atlanta Classification) will be obtained from medical records at hospital discharge. Subsequently, each subject will be prospectively followed at 3 months and 1 year after hospital discharge. In each follow-up, he/she will be asked to answer a questionnaire focusing on symptoms of exocrine pancreatic insufficiency and quality of life. Furthermore, blood and stool samples will be collected at the 3 and 12-month follow up for measurement of nutritional markers and fecal elastase-1 levels.

Based on available literature and our own data, we hypothesize that a significant fraction of AP patients develop EPI that may persist up to 1 year after the discharge, and result in nutritional deficiencies and impaired QOL. This study will help to clarify the incidence, natural history and duration of EPI, as well as identify subgroups of patients at high risk of EPI after AP. It will serve as the basis for the design of future randomized controlled trials of pancreatic enzyme replacement following AP. This is a novel proposal by an investigator with extensive experience and a well-established record in AP research from an internationally known pancreas center of excellence. The methodological strength of our proposal lies on its prospective nature, the 1-year follow up with serial assessments of EPI, nutritional status and QOL, and the detailed phenotypical characterization of the AP patient cohort.

Primary endpoints

* Measure the incidence of exocrine pancreatic insufficiency at 12 months after an attack of AP.

Secondary endpoints

* Identify subgroups of patients at risk for EPI at 12 months after an attack of AP based on severity classification, etiology, and demographics.
* Measure the incidence of transient (present at 3 but no at 12 months) and persistent (present both at 3 and 12 months after AP) exocrine pancreatic insufficiency following an AP attack.
* Measure the incidence of nutritional deficiencies, and impaired quality of life at 3 and 12 months from an attack of AP.
* Assess whether EPI is associated with nutritional deficiencies or impaired quality of life at 3 and 12 months from an AP attack.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, at least 18 years of age, admitted at the University of Pittsburgh Medical Center with an AP attack defined as the presence of 2 or more of the following criteria:

  * Abdominal pain consistent with the disease,
  * Serum amylase and/or lipase greater than three times the upper limit of normal, and or
  * Characteristic findings from abdominal imaging (i.e. demonstrating pancreatic edema, peripancreatic fat stranding or complications or acute pancreatitis)

Exclusion Criteria:

* Known or newly diagnosed chronic pancreatitis based on cross sectional imaging findings
* Pre-existing exocrine pancreatic insufficiency (meaning EPI present before the onset of AP; development of EPI during early refeeding is not an exclusion criterion)
* History of gastric or pancreatic resection
* History of small bowel disease (celiac disease, or Crohn's disease)
* History of pancreatic malignancy
* History of gastroparesis
* History of cystic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women, at least 18 years of age, admitted at the University of Pittsburgh Medical Center with an AP attack defined as the presence of 2 or more of the following criteria:
  * Abdominal pain consistent with the disease,
  * Serum amylase and/or lipase greater than three times the upper limit of normal, and or
  * Characteristic findings from abdominal imaging (i.e. demonstrating pancreatic edema, peripancreatic fat stranding or complications or acute pancreatitis)
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Exocrine pancreatic insufficiency at 12 months | 12 months
  Fecal elastase-1 levels EPI below 200 mcg/g stool,

CONTACTS AND LOCATIONS:
Overall Officials: Georgios I Papachristou, MD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - The Ohio State University, Columbus, Ohio
  - UPMC Presbyterian, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
In the future, the data may be shared with other entities. If so, the research data/documents will be coded and subject identifiers removed prior to access by the external persons.

REFERENCES:
- [Derived] Bejjani J, Culp S, Nikahd M, Phillips AE, Singh V, Roberts KM, Abu-El-Haija M, Krishna SG, Ramsey ML, Lahooti A, Lee PJ, Hart PA, Papachristou GI. Symptom Burden After Acute Pancreatitis and Its Correlation With Exocrine Pancreatic Function: A Multicenter Prospective Study. Clin Transl Gastroenterol. 2025 Feb 1;16(2):e00799. doi: 10.14309/ctg.0000000000000799. PMID 39679584
- [Derived] Phillips AE, Bejjani J, Culp S, Chennat J, Lee PJ, Machicado JD, Singh VK, Afghani E, Ramsey ML, Paragomi P, Stello K, Nikahd M, Hart PA, Papachristou GI. Prevalence of exocrine pancreatic insufficiency at 12 months after acute pancreatitis: a prospective, multicentre, longitudinal cohort study. EClinicalMedicine. 2024 Aug 2;75:102774. doi: 10.1016/j.eclinm.2024.102774. eCollection 2024 Sep. PMID 39210941
- [Derived] Bejjani J, Papachristou GI, Dungan K, Evans Phillips A, Singh V, Toledo FG, Han S, Krishna SG, Lahooti A, Lee PJ, Machicado JD, Nikahd M, Paragomi P, Ramsey M, Yadav D, Culp S, Hart PA. Incident diabetes following acute pancreatitis in a multicenter prospective observational cohort. Pancreatology. 2023 Dec;23(8):900-903. doi: 10.1016/j.pan.2023.10.009. Epub 2023 Oct 10. PMID 37839923
- [Derived] Paragomi P, Phillips AE, Machicado JD, Lahooti A, Kamal A, Afghani E, Pothoulakis I, Reynolds SL, Mays M, Conwell DL, Lara LF, Singh VK, Papachristou GI. Post-Acute Pancreatitis Pancreatic Exocrine Insufficiency: Rationale and Methodology of a Prospective, Observational, Multicenter Cohort Study. Pancreas. 2021 Feb 1;50(2):147-152. doi: 10.1097/MPA.0000000000001743. PMID 33565790